CLINICAL TRIAL: NCT01694030
Title: Effects of Repeated Attachment Security Priming on Depressed Mood: a Clinical Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: University of Southampton: LO6
Record Dates: First submitted 2012-09-17; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Unipolar Depression
Keywords: Attachment security priming; depressed mood
MeSH Terms: conditions — Depressive Disorder; Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neutral Condition (Experimental): Participants in the neutral (control) condition of the attachment security priming experiment will be asked to spend time visualising neutral events (e.g., supermarket shopping)for 3-10 minutes at a time.
  Interventions: Other: Attachment security priming
- Secure condition (Experimental): Participants in the attachment security priming condition will be asked to complete visualisation tasks where they think about a secure attachment figure for between 3 - 10 minutes.
  Interventions: Other: Attachment security priming

INTERVENTIONS:
Other: Attachment security priming

SUMMARY:
The purpose of this study is to explore whether asking participants to visualise a secure attachment figure or a neutral event leads to differences in self-reported felt security or depressed mood. Furthermore, the investigators aim to explore whether it is possible to keep a secure prime activated over 3 days via text message visualisation tasks.

ELIGIBILITY:
Inclusion Criteria:

-Anxiety and depressive symptoms

Exclusion Criteria:

-Bipolar disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Depressed Mood 1 | Depressed mood will be measured on day 7 of the study (immediately after lab primes)
  Depressed mood will be measured using the depression and anxiety items from the Profile of Mood States (POMS: McNair, Lorr, & Droppleman, 1992), which equates to 24 items out of the original 65 on the POMS. Respondents use a 5-point Likert-type scale (0=Not at all, 4=Extremely) to rate the extent to which they have experienced various mood states over the past week. This questionnaire takes 5 minutes to complete.

SECONDARY OUTCOMES:
Felt Security 1 | Felt security will be measured on day 7 of the study (after initial lab primes)
  To find out whether the experimental manipulation was successful, participants will complete a 16-item measure of Felt Security (Luke, Carnelley, & Sedikides, 2012). This scale consists of ten words relating to feelings of security, comfort and safety (e.g., loved, protected). Participants rate the extent to which the person or scenario in the visualisation task made them feel secure, by rating each item using a 6-point Likert-type scale (1=not at all, 6=very much). This measure takes 3 minutes to complete.
Depressed Mood 2 | Depressed mood will be measured on day 7 of the study (after 3 days of text primes)
  Depressed mood will be measured using the depression and anxiety items from the Profile of Mood States (POMS: McNair, Lorr, & Droppleman, 1992), which equates to 24 items out of the original 65 on the POMS. Respondents use a 5-point Likert-type scale (0=Not at all, 4=Extremely) to rate the extent to which they have experienced various mood states over the past week. This questionnaire takes 5 minutes to complete.
Depressed Mood 3 | Depressed mood will be measured on day 11 of the study (24 hours after the last text prime).
  Depressed mood will be measured using the depression and anxiety items from the Profile of Mood States (POMS: McNair, Lorr, & Droppleman, 1992), which equates to 24 items out of the original 65 on the POMS. Respondents use a 5-point Likert-type scale (0=Not at all, 4=Extremely) to rate the extent to which they have experienced various mood states over the past week. This questionnaire takes 5 minutes to complete.
Felt Security 2 | Felt security will be measured on day 10 of the study (after 3 days of text primes)
  Participants will complete a 16-item measure of Felt Security (Luke, Carnelley, & Sedikides, 2012). This scale consists of ten words relating to feelings of security, comfort and safety (e.g., loved, protected). Participants rate the extent to which the person or scenario in the visualisation task made them feel secure, by rating each item using a 6-point Likert-type scale (1=not at all, 6=very much). This measure takes 3 minutes to complete.
Felt Security 3 | Felt security will be measured on day 11 of the study (24 hours after last text prime)
  To find out whether the experimental manipulation was successful, participants will complete a 16-item measure of Felt Security (Luke, Carnelley, & Sedikides, 2012). This scale consists of ten words relating to feelings of security, comfort and safety (e.g., loved, protected). Participants rate the extent to which the person or scenario in the visualisation task made them feel secure, by rating each item using a 6-point Likert-type scale (1=not at all, 6=very much). This measure takes 3 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Baldwin, Principal Investigator — University of Southampton
Locations (1):
- College Keep, Southampton, Hants, United Kingdom